CLINICAL TRIAL: NCT01192711
Title: An Open Label, Multicentre, Randomized Study of Insulin Glargine + Prandial Insulin Glulisine Associated With a Telemedicine System for Carbohydrates Counting vs. Insulin Glargine + Prandial Insulin Glulisine Associated With Common Practice
Brief Title: Insulin Administration Plus a Telemedicine System (Diabetes Interactive Diary - DID) vs Insulin Plus Common Practice
Acronym: DID3
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorzio Mario Negri Sud (Other)
Collaborators: Sanofi (Industry); LifeScan (Industry)
Responsible Party: Antonio Nicolucci/Chair of the Steering Committee, Consorzio Mario Negri Sud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTD003
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2010-09

CONDITIONS: Type 1 Diabetes
Keywords: diabetes; telemedicine; self monitoring blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- insulin + DID (Experimental): Three prandial (before or at the end of meal administration, based on doctor counselling and patient decision) injections per day of insulin glulisine associated with basal insulin glargine; the DID will be used to estimate the CHO content of the food intended to eat. Insulin doses in this group will be adjusted based on DID calculations and pre-meal BG values.
  Interventions: Device: Diabetes Interactive Diary (DID)
- insulin + usual care (No Intervention): Three prandial (before or at the end of meal administration, based on doctor counselling and patient decision) injections of insulin glulisine associated with basal insulin glargine. Insulin doses in group B will be adjusted based on SMBG values reviewed during the doctor office visit.

INTERVENTIONS:
Device: Diabetes Interactive Diary (DID) — DID is both a CHO/insulin bolus calculator, an information technology and a telemedicine system based on the communication between health care professional (physician or dietitian) and patient by SMS messages.
  Arms: insulin + DID

SUMMARY:
The Diabetes Interactive Diary (DID) is both a CHO (carbohydrates )/insulin bolus calculator, an information technology and a telemedicine system based on the communication between health care professional and patient by SMS messages.

Aim of the study is to compare an insulin regimen of insulin glargine + prandial insulin glulisine associated with a telemedicine system to teach CHO counting (DID) with the same insulin regimen administered according to usual practice.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with type 1 diabetes as defined by the criteria of the Expert Committee on the Diagnosis and Classification of Diabetes Mellitus (29)
* Males and females
* Age equal or more than 18 years
* Patients not habitually using CHO (carbohydrates) counting
* Self monitoring blood glucose (SMBG) at least 3 times a day
* Four basal-bolus daily injections of short-acting and long-acting insulin analogues
* HbA1c equal or more than 7.5%
* Female patients have to be postmenopausal, hysterectomised or surgically sterilized or using reliable and adequate contraceptive methods (oral contraception or IUD);
* A full study-specific informed consent must be obtained in writing for all subjects

Exclusion Criteria:

* Multiple daily injections of NPH insulin or soluble rapid insulin or Continuous Subcutaneous Insulin Infusion (CSII) therapy
* Mental conditions, depression, or high anxiety rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Eating disorders
* Pregnancy / lactation.
* Any clinically significant major organ system disease such as relevant cardiovascular, gastrointestinal, hepatic, neurological, endocrine, haematological or other major systemic diseases or infective diseases making implementation of the protocol or interpretation of the study results difficult
* Any disease or condition including abuse of illicit drugs, prescription medicines or alcohol that in the opinion of the investigator may interfere with the completion of the study
* Subjects unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Blood levels of glycosylated hemoglobin | from baseline every three months until the end of the study

SECONDARY OUTCOMES:
blood glucose (BG) levels | from baseline every three months until the end of the study
  Changes in BG levels from baseline to end of study (fasting BG, pre-/post-prandial BG, nocturnal BG, mean daily BG)
Glucose variability | from baseline every three months until the end of the study
  Glucose variability (MAGE, coefficient of variation of mean fasting BG and post-prandial BG)
Change in body weight and BMI | from baseline every three months until the end of the study
Total daily insulin dose, total basal insulin dose, total prandial insulin dose | from baseline every three months until the end of the study
Quality of life | at baseline and at the end of the study
  the quality of life will be measured by Diabetes Specific Quality of Life Scale (DSQOLS) and Diabetes Treatment Satisfaction Questionnaire (DTSQ)
Frequency of patients with hypoglycemic episodes and frequency of hypoglycemic episodes overall | every three months until the end of the study
Frequency of patients with severe and/or symptomatic hypoglycemia and frequency of severe and/or symptomatic hypoglycemic episodes overall | every three months until the end of the study
Frequency and times of hypoglycemic events with regard to occurrence during the day (24 hours) and total treatment duration (24 weeks) | every three months until the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Nicolucci, MD, Study Chair — Consorzio Mario Negri Sud
Locations (13):
- Italy (13):
  - Ospedale G.B. Morgagni - L. Pierantoni, Forlì
  - P.O. di Grosseto - Stabilimento Misericordia, Grosseto
  - Az. Osp. S. Anna - Presidio Ospedaliero Cantù - Mariano Comense, Mariano Comense
  - Istituto Scientifico San Raffaele, Milan
  - Ospedale Niguarda Cà Granda, Milan
  - II Università di Napoli Centro Regionale di Diabetologia Pediatrica "G. Stoppoloni", Naples
  - Università degli Studi di Padova Dipartimento di Medicina Clinica e Sperimentale, Padua
  - Ospedale Cisanello, Pisa
  - U.O. di Diabetologia, Dip. di Malattie Digestive & Metaboliche, Ravenna
  - Ospedale Infermi, Rimini
  - Ospedale Sandro Pertini, Rome
  - Ospedale Magati, Scandiano
  - Azienda Ospedaliera-Universitaria S. Giovanni Battista, Turin